CLINICAL TRIAL: NCT05345704
Title: Simulation-based Comparative Study on Efficiency of Ventilation During Paediatric Cardiopulmonary Resuscitation in Health Care Professionals and Lay Rescuers
Brief Title: Simulation-based Comparative Study on Efficiency of Ventilation During Paediatric Cardiopulmonary Resuscitation
Acronym: PEDIVENT
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Simulation Centre of the Faculty of Medicine of Masaryk University (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: SIMU 2022
Record Dates: First submitted 2022-04-10; First posted 2022-04-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Simulated Pediatric CRP Ventilation
Keywords: CPR; resuscitation; pediatric; ventilation; effectiveness
MeSH Terms: conditions — Respiratory Aspiration | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lay rescuers: Volunteer participants in a role lay rescuers
  Interventions: Other: cardiopulmonary resuscitation (CPR)
- Health care professionals (HCPs): Health care professionals (HCPs) trained in advanced life support
  Interventions: Other: cardiopulmonary resuscitation (CPR)

INTERVENTIONS:
Other: cardiopulmonary resuscitation (CPR) — Data from observation and collected from simulation mannequin during simulated CPR of an infant and child.

SUMMARY:
The aim of this study is to gather data to support beginning the pediatric cardiopulmonary resuscitation (CPR) with 5 initial breaths. The group of health care professionals and the group lay rescuers will be asked to perform cardiopulmonary resuscitation (CRP) on 2 pediatric simulation mannequins (the 3-month-old infant, 5 kg, and the 5-year-old child, 25 kg) and the effectiveness of initial ventilation attempts will be evaluated.

DETAILED DESCRIPTION:
There is a lack of knowledge on the efficiency of ventilation during simulated and real cardiopulmonary resuscitation of children and infants. The ventilations should be an integral part of pediatric resuscitation as recommended by European Resuscitation Council (ERC) because the respiratory and other secondary causes with oxygen depletion are common causes of cardiac arrest in children. However, the effectiveness and quality of ventilation are rarely studied and ERC guidelines to start ventilation with 5 initial breaths in pediatric CPR are based on the experts´ opinion. This study evaluates ventilation efficiency during simulated pediatric cardiopulmonary resuscitation performed by 2 different groups of potential rescuers - physicians, nurses- representing the advanced life support and lay rescuers- representing the basic life support algorithm. The primary aim of this study is to evaluate the number of effective breaths (define as a visible chest rise) during 5 initial breaths attempts of simulated pediatric cardiopulmonary resuscitation. Secondary outcomes include subanalysis of the effectiveness of two initial breaths attempts, defined as a visible chest rise, time to first effective breath, breath volume delivered during 5 initial breaths, and breaths during CPR. The appropriate volume would be considered 6-10 mL/kg (i.e. 30 - 50 mL in infant and 125- 250 mL in the child). The data will be obtained before and after standardized simulation training in both groups. For lay rescuers, the dispatcher-assisted CPR will be simulated. For the health care professionals, basic equipment will be available and expected to be used (correct size mask and bag-mask ventilation).

ELIGIBILITY:
Inclusion Criteria:

* Volunteer participants - lay rescuers
* Health care professionals performing simulated CPR

Exclusion Criteria:

* not willing to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteer participants in a role lay rescuers and Health care professionals (HCPs) trained in advanced life support
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Initial ventilation effectivity | During 90 seconds of life support
  Number of ventilations that are effective out of the first 5 attempts in each group. Defined as breath that has the ability to elevate the chest

SECONDARY OUTCOMES:
Delay in ventilation | During 90 seconds of life support
  Time to first effective ventilation
Initial 2 breaths effectivity | During 90 seconds of life support
  Number of effective ventilation from first 2 ventilation attempts in each group
Initial ventilation adequacy | During 90 seconds of life support
  Number of ventilations with correct volumes (6-8 mL/kg) out of the first 5 attempts
Ventilation volume during initial breaths | During 90 seconds of life support
  Percentage of correct volume breaths during CPR
Delay in CPR | During 90 seconds of life support
  Time to start of chest compressions
CPR description | During 90 seconds of life support
  Number of CPR cycles (15 compressions: 2 ventilations) during 90 seconds of simulated CPR

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided